CLINICAL TRIAL: NCT04213729
Title: A Holistic Diet Intervention for People With Crohn's Disease
Brief Title: Diet Intervention for Crohn's Disease Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Principal Investigator, Maria Abreu, Professor of Medicine, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20190548
Record Dates: First submitted 2019-12-24; First posted 2019-12-30 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Crohn Disease
Keywords: Inflammatory bowel disease (IBD); Diet; CD; IBD; Psychological support; Family member; Low fat, high fiber; Dyadic
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Crohn's Disease (CD) Control Group (Active Comparator): Participants will receive only the one time standard of care in-clinic diet counseling at visit 1.
  Interventions: Behavioral: Diet Counseling
- Experimental CD Low Fat Diet (LFD) Group (Experimental): Participants will be provided catered LFD meals for 8 consecutive weeks consisting of daily breakfast, lunch, dinner and snacks.
  Interventions: Other: CD LFD
- Experimental CD LFD + DPS Group (Experimental): Participants and one family member that lives with them will be provided catered LFD meals for 8 consecutive weeks consisting of daily breakfast, lunch, dinner and snacks. In addition, the participant and their family member will receive 12 consecutive weeks of Dyadic Psychological Support (DPS).
  Interventions: Other: CD LFD; Behavioral: Dyadic Psychological Support (DPS)

INTERVENTIONS:
Behavioral: Diet Counseling — Standard of care diet counseling provided at clinic visit 1.
  Arms: Crohn's Disease (CD) Control Group
Other: CD LFD — Daily breakfast, lunch, dinner and snacks LFD catered meals. Meals will have approximately 20% calories from fat, a goal ratio close to 1:1 omega-6/omega-3 fatty acids, and approximately 25-35 grams of fiber per day.
  Arms: Experimental CD LFD + DPS Group; Experimental CD Low Fat Diet (LFD) Group
Behavioral: Dyadic Psychological Support (DPS) — The dyadic psychosocial support (DPS) intervention will be provided for a total of 12 weeks. The 12-week DPS intervention consists of eight sessions (main sessions) and two booster sessions. The intervention will incorporate psychoeducational components that combine didactic and behavioral regulatory procedures to promote healthy diet behavior for self-determined reasons.
  Arms: Experimental CD LFD + DPS Group

SUMMARY:
The purpose of this study is to determine the effectiveness of a low-fat, high fiber diet (LFD) containing a minimal proportion of fat to improve gastrointestinal symptoms, quality of life and signs of inflammation in blood and stool.

ELIGIBILITY:
Inclusion Criteria for Crohn's disease:

* Male or Female ≥18 and ≤70 years old and lives with someone that is involved in daily diet
* Documented diagnosed of Crohn's Disease
* sCDAI less than 400
* Patients on oral 5-aminosalicylates, mesalamine or sulfasalazine must be on a stable dose for ≥2 weeks prior to screening
* Treated with anti-Tumor Necrotic Factors (TNFs) or immunosuppressants (AZA, 6-Mercaptopurine (6-MP), or methotrexate) at screening must have been on a stable dose for ≥4 weeks
* On steroids can be on no more than prednisone 20 mg daily or budesonide 9 mg daily at the screening. If clinically indicated, tapering of steroids after 4 weeks of intervention may occur. Prednisone may be tapered by no more than 2.5mg/wk and budesonide by no more than 3 mg/wk.
* No antibiotic use or probiotic use within 2 weeks prior to screening

Exclusion Criteria for Crohn's disease:

Patients with Ulcerative Colitis and Celiac Disease

* Abdominal abscess, symptomatic Intestinal stricture, patients with altered anatomy: prior total colectomy or proctocolectomy or anticipated colectomy during the study period and presence of ileal pouch or ostomy
* Other clinically meaningful laboratory abnormalities: pregnancy or lactation, an unstable or uncontrolled medical disorder, colonic dysplasia or adenomas, and malignant neoplasms. Toxic megacolon situations such as Patients with short life expectancy
* Use of cyclosporine, mycophenolate mofetil, sirolimus, thalidomide or tacrolimus within 2 months prior to screening
* Need for prednisone > 20 mg daily or budesonide > 9 mg daily at the time of screening. Received intravenous corticosteroids within 2 weeks prior to screening, during screening, or during the study period except as premedication for anti-TNFs
* Use of Total Parenteral Nutrition at the time of screening and during the study period.
* Presence of any of the following laboratory abnormalities during screening period or at least <12 weeks; Hemoglobin <8.0g/dl, Albumin <2.8g/dl.
* Uncooperative behavior or any condition that could make the patient potentially noncompliant to the study procedure
* Other significant or life-threatening co-morbidities in which low fat/high fiber diet intervention could negatively affect
* The need for antibiotic use during the study period
* Known allergy to tree nuts or peanuts
* Pregnant women

Inclusion and Exclusion Criteria for Family-like Member

Inclusion:

* Male or Female ≥18 and ≤70 years old
* Live in the same household and be involved in the patients' daily diet
* No antibiotic use or probiotic use within 2 weeks prior to screening

Exclusion Criteria

* Patients with Ulcerative Colitis and Celiac Disease
* Abdominal abscess, symptomatic Intestinal stricture, patients with altered anatomy: prior total colectomy or proctocolectomy or anticipated colectomy during the study period and presence of ileal pouch or ostomy
* Other clinically meaningful laboratory abnormalities: pregnancy or lactation, an unstable or uncontrolled medical disorder, colonic dysplasia or adenomas, and malignant neoplasms. Toxic megacolon situations such Uncooperative behavior or any condition that could make the patient potentially noncompliant to the study procedures. Patients with short life expectancy
* Use of cyclosporine, mycophenolate mofetil, sirolimus, thalidomide or tacrolimus within 2 months prior to screening
* Use of Total Parenteral Nutrition at the time of screening and during the study period.
* Other significant or life-threatening co-morbidities in which low fat/high fiber diet intervention could negatively affect
* The need for antibiotic use during the study period
* Known allergy to tree nuts or peanuts
* Pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Change in fat intake | Baseline, 8 weeks
  Change in daily fat intake calculated through patient reported diet diary app Nutrihand.
Rate of adherence to fat intake | Week 36
  Adherence to fat intake is measured by the web-based Automated Self-Administered 24-hour diet recall (ASA24).

SECONDARY OUTCOMES:
Change in clinical symptoms as assessed by Patient Reported Outcomes (PRO2). | Baseline, Week 8
  PRO2 is the sum of the average daily stool frequency and abdominal pain. A weighted total PRO2 score of less than 75 is an indication of remission.
Change in clinical symptoms as assessed by the Harvey Bradshaw Index (HBI) | Baseline, Week 8
  HBI is a 5-item questionnaire. An HBI score of <5 indicates remission, 5-7 indicates mild disease, 8-16 indicates moderate disease and >16 indicates severe disease.
Change in clinical symptoms as assessed by the Short Crohn's Disease Activity Index (sCDAI). | Baseline, Week 8
  sCDAI is the sum of the average daily stool frequency, general well-being and abdominal pain. A weighted total sCDAI score of less than 150 indicates remission, 150-219 indicates mild activity, 220-450 indicates moderate activity and > 450 indicates severe activity.
Change in quality of life (QoL) as assessed by the Short Inflammation Bowel Disease Questionnaire (sIBDQ). | Baseline, Week 8
  sIBDQ is a 10-item shortened version of the original IBDQ assessing QOL with total scores ranging from 1 to 7 with a higher score indicating a better QOL.
Change in quality of life (QoL) as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS-29). | Baseline, Week 8
  The PROMIS-29, a generic health-related quality of life survey, assesses each of the 7 PROMIS domains with 4 questions. The questions are ranked on a 5-point Likert Scale. There is also one 11-point rating scale for pain intensity. A score of 50 represents the mean or average of the reference population. A score of 60 means that the person is one standard deviation above the reference population (standard deviation = 10).
Change in the expression of cytokine high-sensitivity C-reactive protein (hsCRP). | Baseline, Week 8
  Change in the expression of cytokine high-sensitivity C-reactive protein (hsCRP) evaluated in mg/L.
Change in the expression of Serum Amyloid A (SAA). | Baseline, Week 8
  Change in the expression of SAA evaluated in pg/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Maria T Abreu, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No